CLINICAL TRIAL: NCT03832725
Title: Pathobiology of Remission of Type 2 Diabetes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Tennessee (Other)
Responsible Party: Principal Investigator, Frankie Stentz, Professor/ Department of Medicine/Endocrinology, Diabetes and Metabolism, University of Tennessee
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: UTennHSCFS
Record Dates: First submitted 2019-02-01; First posted 2019-02-06 (Actual); Last update posted 2019-02-07 (Actual); Status verified 2019-02

CONDITIONS: Newly Diagnosed Type 2 Diabetes; Obese
Keywords: Type 2 Diabetes; obesity; pathobiology
MeSH Terms: conditions — Obesity; Diabetes Mellitus, Type 2 | interventions — Diet, Reducing

STUDY DESIGN:
Intervention Model Description: Subjects will be randomized to a macronutrient high protein or high carbohydrate diet provided by the study for weight loss and remission of Type 2 Diabetes
Who Masked: Participant, Investigator
Masking Description: Subjects or investigators will not know which macronutrient diet (high protein or high carbohydrate) which they are given for the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High protein (HP) weight loss diet (Active Comparator): A weight loss high protein (HP) (30% Kcal protein, 40% Kcal carbohydrate (CHO) and 30% Kcal fat) diet will be given to the subjects on that arm of study to pick up weekly for 6 months.
  Interventions: Other: High Protein (HP) weight loss diet
- High carbohydrate (HC) weight loss diet (Active Comparator): A weight loss high carbohydrate (HC) (15% Kcal protein, 55% Kcal CHO and 30% Kcal fat) diet will be given to the subjects on that arm of study to pick up weekly for 6 months.
  Intervention with the HC diet will be 6 months. If subjects have not had remission of Type 2 Diabetes by the end of the 6 months, they will be referred to an endocrinologist for pharmaceutical treatment
  Interventions: Other: High carbohydrate (HC) weight loss diet

INTERVENTIONS:
Other: High Protein (HP) weight loss diet — Newly diagnosed Type 2 Diabetic (NT2DM) subjects will be placed on a HP diet for 6 months with all food provided for weight loss and remission of NT2DM.
  Intervention with the HP diet will be 6 months. If subjects have not had remission of Type 2 Diabetes by the end of the 6 months, they will be referred to an endocrinologist for pharmaceutical treatment
  Arms: High protein (HP) weight loss diet
Other: High carbohydrate (HC) weight loss diet — Newly diagnosed Type 2 Diabetic (NT2DM) subjects will be placed on a HC diet for 6 months with all food provided for weight loss and remission of NT2DM.
  Intervention with the HP diet will be 6 months. If subjects have not had remission of Type 2 Diabetes by the end of the 6 months, they will be referred to an endocrinologist for pharmaceutical treatment
  Arms: High carbohydrate (HC) weight loss diet

SUMMARY:
We propose to investigate effects of HP and HC weight loss diets in Newly Diagnosed T2DM (NT2DM) women and men for 6 months for remission of Type 2 Diabetes. Our long term goal is to establish a weight loss diet plan for remission of NT2DM which would be adaptable for use in physicians' clinics and metabolomics predictors for assessment of remission. The overall objective of this study is to determine if remission of NT2DM can be induced by dietary manipulation using a HP diet and the pathobiology of this remission. We hypothesize that NT2DM subjects will have remission to NGT on the HP diet when they are provided the food and daily menus for compliance. The rationale is the HP diet is palatable for subjects to continue after the 6 month study and stay in remission using diet plans we provide. We will compare the effects of the HP vs HC diet on remission. Specific aims of this study are to determine the effects of the HP and HC diets on NT2DM obese subjects in a 6 month feeding study and determine: (a)remission of NT2DM to Normal Glucose Tolerance(NGT), (b)weight loss, (c)improvements in metabolic markers, Cardiovascular Risk Factors(CVR), and inflammation markers, and epigenetic DNA methylation changes and pathways involved with remission and metabolomic markers to establish predictive markers of remission of NT2DM. We propose to use a non-pharmaceutical means (HP diet) for remission of T2DM and weight loss and determine the pathobiology involved in improvement in metabolic and CVRs by interrogating the samples with emerging technologies. The proposed research is significant because if we can demonstrate the HP diet cause remission of NT2DM to NGT along with other metabolic improvements, it would be a significant improvement in health risk and medical cost to subjects.

DETAILED DESCRIPTION:
Greater than 30 million people have diabetes. Over time diabetic patients need more and more medications and develop numerous medical complications. Remission of Type 2 Diabetes (T2DM) would have profound effects on people with diabetes with respect to overall health improvement (insulin sensitivity(Si), cardiovascular risk factors(CVR), inflammation markers (IC)), reduction of retinopathy, nephropathy, neuropathy and reduction in medical costs. Methods to accomplish this have not yet been determined, however, it is generally accepted that non-drug methods to treat T2DM is the most cost effective and have the fewest side effects. The primary risk factor for T2DM is obesity. Our randomized clinical trials comparing the effects of High Protein (HP) vs High Carbohydrate (HC) weight loss diets in obese, prediabetic(IGT) women and men where all foods were provided daily for 6 months(mo) showed that while both diet groups had similar weight loss, 100% of HP diet subjects had remission from IGT to Normal Glucose Tolerance(NGT), but only 33% of HC diet group had remission. Also, the HP diet provided greater improvement in Si, CVR, IC, and an increase in % lean body mass (LBM) compared to the HC diet demonstrating that weight loss is not the only factor involved in remission. Based on these findings, we now propose to investigate effects of HP and HC weight loss diets in Newly Diagnosed T2DM (NT2DM) women and men for 6 mo. Our long term goal is to establish a weight loss diet plan for remission of NT2DM which would be adaptable for use in physicians' clinics and metabolomics predictors for assess-ment of remission. The overall objective of this study is to determine if remission of NT2DM can be induced by dietary manipulation using a HP diet and the pathobiology of this remission. We hypothesize that NT2DM subjects will have remission to NGT on the HP diet when they are provided the food and daily menus for compliance. The rationale is the HP diet is palatable for subjects to continue after the 6 mo study and stay in remission using diet plans we provide. We will compare the effects of the HP vs HC diet on remission. Specific aims of this study are to determine the effects of the HP and HC diets on NT2DM obese subjects in a 6 mo feeding study and determine: (a)remission of NT2DM to NGT, (b)weight loss and LBM preservation, (c)improvements in metabolic markers, CVRs, IC, epigenetic DNA methylation changes and pathways involved with remission and metabolomic markers to establish predictive markers of remission of NT2DM. This study is innovative in that we propose to use a non-pharmaceutical means (HP diet) for remission of T2DM diabetes and weight loss and determine the pathobiology involved in improvement in metabolic and CVRs by interrogating the samples with emerging technologies. The proposed research is significant because if we can demonstrate the HP diet cause remission of NT2DM to NGT along with other metabolic improvements, it would be a significant improvement in health risk and medical cost to subjects

ELIGIBILITY:
Inclusion Criteria:

i) Age range 20 yrs to 50 yrs; ii) BMI > 30 kg/m2 to 55kg/m2; iii). Fasting blood glucose >126 mg/dl and 2 hour glucose >200 mg/dl determined by OGTT; iv). HbA1c > 6.5 % to ≤10%.

-

Exclusion Criteria:

i) Proteinuria or elevated serum creatinine (>1.5 mg/dl); ii) Surgical or premature menopause; iii) liver disease or abnormal liver function tests; iv) T2DM of greater than 2 yrs; v) Thyroid disease with abnormal TSH; vi) Weight > 350 lbs, (due to fit on DXA); vii) Triglycerides>400 mg/dl or LDL cholesterol >160 mg/dl; viii) SBP>145, DBP>100 mm of Hg; ix) on medications known to effect lipid or glucose metabolism; x) Pregnancy or become pregnant in next 6 mo; xi) Weight loss >10% of body weight in last 6 mo; xii)History of cancer <5 yrs or undergoing active treatment; xiii) smoking, xiv)alcohol abuse; xv) having CPAP treatment. xvi)Subjects with HbA1c >10% will be referred to an endocrinologist for pharmacological treatment.

-

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2018-03-01 (Actual); Primary Completion 2024-07-31 (Estimated); Study Completion 2024-07-31 (Estimated)

PRIMARY OUTCOMES:
Remission of Type 2 Diabetes | Each subject will be monitored for 6 months while they are on the HP or HC diet for remission of Type 2 Diabetes
  Remission of NT2DM to NGT will be determined by the OGTT ( a 75 gm glucose drink given at 0 minutes and then blood drawn to determine the glucose level at 2 hrs). This OGTT will be done at 3 and 6 months with the criteria of fasting glucose <126 mg/l and 2 hour glucose <140 mg/dl. Criteria for improvement from NT2DM to IGT will be fasting blood glucose <126 mg/dl and 2 hour glucose <199 mg/dl. At each weekly visit for food pick up the subject's glucose will be monitored for blood glucose changes from the start of the diet study. If subjects do not have remission of diabetes at 6 months, they will be referred to an endocrinologist for possible pharmacology treatment.

SECONDARY OUTCOMES:
Weight loss | Each subject will be monitored for 6 months while they are on the HP or HC diet
  Determine changes in weight loss changes in inflammation markers such as cytokines, changes in incretins and determine metabolom markers for diagnosis of remission of NT2DM over the 6 months of the study
Cardiovascular Risk Factors (CVR) | Each subject will be monitored for 6 months while they are on the HP or HC diet
  Changes in CVR will be determined by changes in blood pressure (systolic/diastolic) from the start of the diet to the end of the 6 month diet study.
Inflammation markers such as cytokines, | Each subject will be monitored for 6 months while they are on the HP or HC diet
  Changes in inflammation markers in the subjects' blood such as cytokines
Metabolom Markers | Each subject will be monitored for 6 months while they are on the HP or HC diet
  Changes in Metabolom Markers will be measured to determine changes from the start of the study to the end of the 6 months for possible markers of remission diabetes

CONTACTS AND LOCATIONS:
Overall Officials: Frankie B Stentz, PhD, Principal Investigator — University of Tennessee
Locations (1):
- University of Tennessee Health Science Center, Memphis, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Yes
Study protocol and informed consent will be shared. Data at the end of the study will be reported. No patient identification will be shared.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Over the time frame of the study
Access Criteria: contact investigator